CLINICAL TRIAL: NCT06725758
Title: A Phase 1/2, First-in-Human Study On ODM-212 In Subjects With Selected Advanced Solid Tumours
Acronym: TEADES
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3134001; 2022-503061-29-00 (EU CTIS Number); U1111-1291-5455 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2024-11-29; First posted 2024-12-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumours
Keywords: Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ODM-212 (Experimental): ODM-212 5mg and/or 40mg tablets
  Interventions: Drug: ODM-212

INTERVENTIONS:
Drug: ODM-212 — ODM-212 5mg and/or 40mg tablets

SUMMARY:
Multi-site, open-label, first-in-human study with 2 parts (dose escalation and dose expansion) in subjects with selected advanced solid tumours

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years old
2. Subjects must have histological diagnosis of locally advanced (primary or recurrent) or metastatic solid tumour of the kind listed below that is not amenable for treatment with curative intent, e.g.:

   Part 1:
   * mesothelioma
   * epithelioid hemangioendothelioma (EHE)
   * cholangiocarcinoma (CCA)
   * head and neck squamous cell carcinoma (HNSCC)
   * non-small cell lung carcinoma (NSCLC)
   * colorectal cancer (CRC)
   * hepatocellular cancer (HCC)
   * castration-resistant prostate cancer (CRPC)
   * meningioma
   * any other solid tumours with available local data for loss-of-function genetic alterations (truncating mutations or gene deletion) in neurofibrin 2 (NF2)/large tumour suppressor kinase (LATS1/LATS2), or Yes-associated protein/ Transiptional coactivator with PDZ-binding motif (YAP/TAZ) fusions
   * any other solid tumour based on emerging scientific data as per sponsor's decision.

   Part 2: Any solid tumour type harbouring a Hippo pathway alteration and other tumour types potentially responsive to transcriptional enhanced associate domain (TEAD) inhibition based on data from Part 1 or other existing or emerging scientific data.
3. Subjects must be in need of systemic treatment for their cancer and to either be refractory to or have progressed on, are intolerant to, or are not otherwise a candidate, in the opinion of the investigator, for any of the currently available established therapies (reasons of unsuitability of standard of care treatments to be recorded).
4. Part 2 only: Subjects must have measurable disease by response evaluation criteria in solid tumours (response evaluation criteria in solid tumors - RECIST) v. 1.1 (modified RECIST for malignant pleural mesothelioma - MPM).
5. Part 2 only: A fresh or recent (taken up to 1 year ago) primary tumour tissue sample from a diagnostic biopsy/surgery or a tumour biopsy taken from a metastasis must be available; exemptions possible by the sponsor's decision.
6. Performance status 0-1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
7. Life expectancy of >12 weeks.
8. Willing and able to comply with all aspects of the protocol.
9. Provide written informed consent (IC; or witness consent) prior to any study-specific screening procedures.

Exclusion Criteria:

1. Other malignancy active within the previous 2 years except for basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast, for which the subject has completed curative therapy.
2. Prior chemotherapy, immunotherapy (tumour vaccine, cytokine or growth factor given to control the cancer) or other anti-cancer therapy within less than 2 weeks before study drug administration, or any persistent unresolved toxicity from previous anti-cancer therapies of common terminology criteria for adverse events (CTCAE) Grade ≥ 2 (except for peripheral neuropathy, alopecia, endocrine disorders that are controlled with replacement hormone therapy and asymptomatic laboratory abnormalities). Especially, care should be exercised to exclude subjects with potential carry-over nephrotoxic effects from previous therapies (e.g., cisplatin). Luteinizing hormone releasing hormone (LHRH) agonists or antagonists are allowed as concomitant treatment.
3. Prior definitive radiation therapy within less than 4 weeks and prior palliative radiotherapy within less than 2 weeks before study drug administration. Radiopharmaceuticals (strontium, samarium) within less than 8 weeks before study drug administration.
4. Subjects with brain or subdural metastases are not eligible, unless the metastases are asymptomatic and do not require treatment or have been adequately treated with local therapy.
5. Known human immunodeficiency virus (HIV) infection.
6. Active infection requiring therapy, including known positive tests for Hepatitis B surface antigen and hepatitis C virus (HCV) Ribonucleic acid (RNA). Pre-study testing for these pathogens is not required.
7. Major surgery within 4 weeks before the first dose of study drug or minor surgery within 1 week (subject must also have recovered from any surgery-related toxicities to less than CTCAE Grade 2).
8. Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (doses >10 mg/day prednisone or equivalent) within 2 weeks before study drug administration.
9. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g. nausea, diarrhoea, or vomiting) that might impair the bioavailability of ODM-212.
10. Use of other investigational medicinal products within 2 weeks or at least5 half-lives (whichever is longer) before study drug administration, or any persistent unresolved toxicity from such treatment that, according to the judgement of the investigator, may pose a health risk for the subject, if taking part in the study. For drugs such as investigational monoclonal antibodies with half-lives >10 days, at least 8 weeks is required. In addition, all visits (apart from survival follow-up) related to the use of another IMP must be completed before dosing with ODM-212 may commence.
11. Use of any live or live-attenuated vaccines (e.g., intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines) within 28 days prior to the first dose of study drug.
12. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG; e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 ms, a prolonged QTc interval (QTcF/B >470 ms) as demonstrated by 2 out of 3 repeated ECG at screening, performed according to local practice. A history of risk factors for torsade de pointes (e.g. heart failure, hypokalaemia, family history of long QT Syndrome) or the use of concomitant medications that prolong the QTc interval.
13. Significant cardiovascular impairment: history of congestive heart failure of New York Heart Association (NYHA) Class III-IV, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke, left ventricular ejection fraction (LVEF) <50%, cardiac arrhythmia requiring medical treatment (including oral anticoagulation) within 6 months prior to the first dose of study drug.
14. Female subjects who are breastfeeding or pregnant at screening or baseline.
15. A separate baseline assessment for pregnancy is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
16. Female subjects of childbearing potential who meet any of the following criteria:

    Had unprotected sexual intercourse within 30 days before study entry or who do not agree to use a highly effective method of contraception (e.g., true abstinence if it is their preferred and usual lifestyle [defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment], an intrauterine device, a contraceptive implant, an oral contraceptive combined with a double barrier method [e.g. combination of male condom with either cap, diaphragm or sponge with spermicide], or have a vasectomized partner with confirmed azoospermia) throughout the entire treatment period and for 28 days after treatment discontinuation.

    Are neither using a highly effective method of contraception (as listed above) nor currently abstinent, or do not agree to refrain from sexual activity during the treatment period and for 28 days after treatment discontinuation.

    Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study and for 28 days after treatment discontinuation.
17. Male subjects who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the treatment period and for 28 days after treatment discontinuation).
18. Urine albumin/creatinine ratio ≥3 mg/mmol (category A2 urine albumin/creatinine ratio [UACR] or higher) in laboratory testing at screening, end-stage renal disease (subjects with eGFR <15 ml/min/1.73 m2, subjects on dialysis and kidney transplant recipients), moderately or severely impaired kidney function (eGFR 15-60 ml/min/1.73 m2), or any pre-existing condition associated with kidney impairment (e.g. subjects with type 1 or type 2 diabetes mellitus and confirmed nephropathy).
19. Hepatic impairment defined as having any of the following laboratory values at screening: total bilirubin ≥1.5xupper limit of normal (ULN) (or >3xULN for subjects with Gilbert's syndrome), aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥3xULN (or ≥5xULN for subjects with liver metastasis), or albumin ≤30 g/L.
20. Abnormalities in coagulation values defined as International Normalised ratio (INR) >1.5xULN at screening (unless subject is receiving anticoagulant therapy, as long as subject's laboratory values are within therapeutic range of intended use of anticoagulants).
21. Haemoglobin <10 g/dL (in absence of blood transfusion within 7 days of value obtained), absolute neutrophil count <1500/µl (1.5 x 109/l), platelet count <100 000/µl (100 x 109/l).
22. Any other major illness, any history of a medical condition or a concomitant medical condition that, in the investigator's judgment, will substantially increase the risk associated with, or compromise the subject's participation in this study.
23. History of treatment with other TEAD inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and frequency of treatment emergent adverse events (TEAE) | From first dose to 1 year after LSLV
  A TEAE is defined as any event arising or worsening after the start of treatment administration until 28 days after the last treatment intake.
Severity of TEAE | From first dose to 1 year after LSLV
  All AEs (except proteinuria which is to be graded according to urine albumin/creatinine ratio (UACR) category) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Royal Marsden Hospital, London, UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No